CLINICAL TRIAL: NCT04116216
Title: Effects of rTMS Associated to Physical Therapy on Motor Function of Parkinson's Disease Patients With Different Phenotypes
Brief Title: rTMS on Motor Function of Parkinson's Disease Patients With Different Phenotypes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Clinical professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMS_PD_phenotype
Record Dates: First submitted 2019-09-23; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High frequency rTMS + physical therapy (Active Comparator): The sessions will be performed five times a week for two weeks. The individuals will be performed the following protocol: first the coil center will be positioned over Cz for the first 1000 pulses. Then the coil will be moved to C4 and C3, where 1000 pulses will be delivered to each hemisphere. The intensity will be set to 100% of the motor threshold. The high frequency stimulation will be delivered at 10 Hz, offered in 20 50-pulse trains, with 30-second train intervals. After rTMS, patients will be submitted to 40 minutes of physical therapy protocol.
  Interventions: Combination Product: High frequency repetitive transcranial magnetic stimulation
- Low frequency rTMS + physical therapy (Active Comparator): The sessions will be performed five times a week for two weeks. The individuals will be performed the following protocol: first the coil center will be positioned over Cz for the first 1000 pulses. Then the coil will be moved to C4 and C3, where 1000 pulses will be delivered to each hemisphere. The intensity will be set to 100% of the motor threshold. The low frequency will be performed at 1 Hz. After rTMS, patients will be submitted to 40 minutes of physical therapy protocol.
  Interventions: Combination Product: Low frequency repetitive transcranial magnetic stimulation
- Sham rTMS + physical therapy (Sham Comparator): For sham stimulation, the stimulator positioned behind the patient will be turned off immediately after the determination of RMT, however, the coil will remain positioned over the patient's scalp (Cz, C3 and C4). A computer equipped with speakers will play an audio recording with the characteristic rTMS sound and no stimulation will be induced in the brain.
  Interventions: Combination Product: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Combination Product: High frequency repetitive transcranial magnetic stimulation — The sessions will be performed five times a week for two weeks. The individuals will be performed the following protocol: first the coil center will be positioned over Cz for the first 1000 pulses. Then the coil will be moved to C4 and C3, where 1000 pulses will be delivered to each hemisphere. The intensity will be set to 100% of the motor threshold. The high frequency stimulation will be delivered at 10 Hz, offered in 20 50-pulse trains, with 30-second train intervals. The low frequency will be performed at 1 Hz. After rTMS, patients will be submitted to 40 minutes of physical therapy protocol.
  Arms: High frequency rTMS + physical therapy
Combination Product: Low frequency repetitive transcranial magnetic stimulation — The sessions will be performed five times a week for two weeks. The individuals will be performed the following protocol: first the coil center will be positioned over Cz for the first 1000 pulses. Then the coil will be moved to C4 and C3, where 1000 pulses will be delivered to each hemisphere. The intensity will be set to 100% of the motor threshold. The high frequency stimulation will be delivered at 10 Hz, offered in 20 50-pulse trains, with 30-second train intervals. The low frequency will be performed at 1 Hz. After rTMS, patients will be submitted to 40 minutes of physical therapy protocol.
  Arms: Low frequency rTMS + physical therapy
Combination Product: Sham repetitive transcranial magnetic stimulation — For sham stimulation, the stimulator positioned behind the patient will be turned off immediately after the determination of RMT, however, the coil will remain positioned over the patient's scalp (Cz, C3 and C4). A computer equipped with speakers will play an audio recording with the characteristic rTMS sound and no stimulation will be induced in the brain.
  Arms: Sham rTMS + physical therapy

SUMMARY:
In this study we wondered whether patients with different phenotypes of Parkinson's disease respond differently to the protocol of repetitive transcranial magnetic stimulation (rTMS) associated with physical therapy. Furthermore, the study aims to compare the effects of rTMS protocols (high and low frequency) associated with physical therapy in PD patients with different phenotypes regarding to motor performance; bradykinesia; functional mobility; balance; quality of life; perception of improvement.

DETAILED DESCRIPTION:
After given prior informed consent, volunteers will be classified and randomized using a website (randomization.com) by a non-involved researcher. At study beginning, volunteers will be evaluated through structured questionnaire. They will be submitted to the following evaluations: (i) Unified Parkinson's disease Rating Scale (UPDRS); (ii) Parkinson's disease Sleep Scale; (iii) Parkinson's disease questionnaire; (iv) Short version of Balance Evaluation Systems Test; (v) Timed up and go; (vi) 5-times sit to stand test; (iv) Patient Global Impression of Change Scale. The cortical activity of the patients will be assessed through electroencephalography and transcranial magnetic stimulation.

Treatment - Participants will be randomly allocated to one of the following experimental protocols: (i) real high frequency rTMS + physical therapy protocol; (ii) real low frequency rTMS + physical therapy protocol; (iii) rTMS sham + physiotherapeutic protocol. The sessions will be performed five times a week for two weeks. Individuals allocated to the high frequency rTMS group will be performed the following protocol: first the coil center will be positioned over Cz for the first 1000 pulses. Then the coil will be moved to C4 and C3, where 1000 pulses will be delivered to each hemisphere. The intensity will be set to 100% of the motor threshold. The high frequency stimulation will be delivered at 10 Hz, offered in 20 50-pulse trains, with 30-second train intervals. The low frequency will be performed at 1 Hz. All groups will be treated with physical therapy immediately after rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PD provided by neurologist;
* Aged 40 or over, of both gender;
* Regular antiparkinsonian pharmacological treatment;
* With staging from I to IV on the modified Hoehn & Yahr scale.

Exclusion Criteria:

* Prior neurological diseases
* Metal implant in the skull and face
* Pacemaker
* History of seizures
* Epilepsy
* Pregnancy
* Other disorders that affect the performance of the tests and proposed intervention
* Other osteomioarticular diseases in the lower limbs that interfere with performance and locomotion
* Submitted to previous surgical intervention for PD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Unified Parkinson's disease Rating Scale - Session III | baseline, after 7 days, after 15 days
  In the present study we will analyze the UPDRS session III which comprises 14 items with a score of 0-4 each, from best to worst motor performance (SHULMAN et al., 2010). According to UPDRS scores, patients will be classified as: (i) tremor-dominant (TD) or (ii) with postural instability and difficulty in walking (PIGD).

SECONDARY OUTCOMES:
Changes on cortical excitability level | baseline, after 7 days, after 15 days
  it will be evaluated through single pulse transcranial magnetic stimulation. Initially, rest motor threshold (RMT) will be determined by finding the lowest stimulator output that elicit motor evoked potential (MEP) around 50 μV (TMS Motor Threshold Assessment Tool -MTAT 2.0 - USA For RMT measure, a figure-eight coil connected to the magnetic stimulator held manually at 45 degrees from the midline, will be placed over the primary motor cortex of most and less impaired hemisphere (C3 and C4 - 10/20 System).
Changes on quality of life | baseline, after 15 days
  It will be evaluated through the score of each domain of Parkinson Disease Questionnaire (PDQ-39), a specific questionnaire for Parkinson's disease. It comprises 39 questions that assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living. Higher values represent a worse perception of quality of life.
Changes on Patient Global Impression of Change Scale | after 15 days
  The PGICS is a one-dimensional measure in which individuals rate their improvement associated with intervention on a scale of 7 items ranging from "1 = no change" to "7 = Much better".

OTHER OUTCOMES:
Changes on balance | baseline, after 15 days
  It will be evaluated by the short version of the Balance Evaluation Systems Test. This test is comprised of 14 full version items that assess the static and dynamic balance of individuals.
Changes on functional mobility to sit-to-stand | baseline, baseline, after 7 days, after 15 days
  It will be assessed through the time of execution during 5-times sit to stand test. The mean of three trials will be recorded to measure fuctional mobility.
Changes on functional mobility | baseline, baseline, after 7 days, after 15 days
  It will be assessed through the time of execution during timed up and go test. The mean of three trials will be recorded to measure fuctional mobility.
Changes on Unified Parkinson's disease rating scale - session II | baseline, baseline, after 7 days, after 15 days
  The total score of this scale will also be used to assess the severity of the disease regarding the performance of daily life activities. The scale ranges a score from 0 to 4 for each question, from best to worst performance.
Changes on sleep quality | baseline, baseline, after 7 days, after 15 days
  Through the Parkinson's Disease Sleep Scale (PDSS), consisting of 15 questions that assesses nocturnal disorders due to PD. Total scores less than 82 or less than five in each sub-item may be indicative of impairment in sleep quality.
Changes on cortical activity | baseline, baseline, after 7 days, after 15 days
  The EEG electrodes will be positioned over the scalp of the patient, according to international marking system 10-20. During the acquisition of the electroencephalographic signal, a protocol (six minutes) of execution and motor imagination will be performed. The collected data will be further processed and analyzed using the MATLAB® software for Windows

CONTACTS AND LOCATIONS:
Overall Officials: Kátia M Silva, PhD, Study Chair — Universidade Federal de Pernambuco
Locations (1):
- Applied Neuroscience Laboratory, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No